CLINICAL TRIAL: NCT06604156
Title: The Effect of the Nociception Index (qNOX) in Painless Gastrointestinal Endoscopy :a Clinical Study
Brief Title: Anesthesia Induction Scheme for Painless Gastrointestinal Endoscopy Patients Based on Nociceptive Stimulation Monitoring
Status: Recruiting | Type: Observational
Sponsor: Min Su (Other)
Responsible Party: Sponsor-Investigator, Min Su, Professor of Anesthesiology, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2024-239-01
Record Dates: First submitted 2024-04-11; First posted 2024-09-19 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Depth of Anesthesia; Nociception; Painless Gastrointestinal Endoscopy
Keywords: Painless Gastrointestinal endoscopy; depth of anesthesia; nociception

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastroscopy group: This study used an EEG bispectral index monitor (Apolo 9000A) to monitor quantitative consciousness (qCON) index and quantitative nociceptive (qNOX) index during gastroscopy. Anesthesia induction was performed using 1.5-2.5mg/kg propofol and 3-5 μ g sufentanil; The injection speed of propofol is between 120s and 180s. When the patient's consciousness disappears (the patient's eyelash reflex disappears, and there is no response to calls and external stimuli), and the Modified Alertness/Sedation (MOAAS) score is ≤ 1, gastroscopy examination will begin. During the examination, propofol 4-12mg/kg. h will be pumped to make MOAA/S ≤ 1, and there will be no body movement reaction.
  Interventions: Device: EEG monitoring
- Colonoscopy group: This study used an EEG bispectral index monitor (Apolo 9000A) to monitor quantitative consciousness (qCON) index and quantitative nociceptive (qNOX) index during Colonoscopy. Anesthesia induction was performed using 1.5-2.5mg/kg propofol and 3-5 μ g sufentanil; The injection speed of propofol is between 120s and 180s. When the patient's consciousness disappears (the patient's eyelash reflex disappears, and there is no response to calls and external stimuli), and the Modified Alertness/Sedation (MOAAS) score is ≤ 1, Colonoscopy examination will begin. During the examination, propofol 4-12mg/kg. h will be pumped to make MOAA/S ≤ 1, and there will be no body movement reaction.
  Interventions: Device: EEG monitoring

INTERVENTIONS:
Device: EEG monitoring — During gastrointestinal endoscopy, electroencephalogram (EEG) monitoring will be conducted using qCON and qNOX technologies to assess patients' sedation and analgesia status while they undergo painless gastrointestinal endoscopy. This will be combined with visual assessments (such as cough reflex, respiratory depression, and limb movement) and clinical physiological monitoring (including vital signs and pulse oximetry) to explore and establish a stable and optimal depth of sedation for anesthesia.

SUMMARY:
Nociception is the encoding and processing of noxious stimulation and is considered an objective indicator for monitoring pain. Currently, a new clinically-applied medical-engineering integrated monitoring device for noxious stimulation response has emerged. Its fundamental principle is based on the monitoring of electroencephalographic (EEG) activity, incorporating two monitoring parameters: the quantitative consciousness (qCON) index and the quantitative nociceptive (qNOX) index. However, in the context of sedation for gastrointestinal endoscopy, how the dynamic changes of the quantitative consciousness index (qCON) and the quantitative nociception index (qNOX) reflect the depth of sedation and nociceptive response remains unclear. Safe and effective sedation monitoring includes both direct visual monitoring and physiological monitoring, that is, monitoring the patient's hemodynamics and depth of sedation. This study utilizes qCON and qNOX monitoring to assess the sedation and analgesic states of patients undergoing painless gastroenterological endoscopy. By combining visual assessment (cough reflex, respiratory depression, and limb movement) with clinical physiological monitoring (vital signs monitoring and pulse oximetry), the aim is to explore the optimal sedation range for gastrointestinal endoscopy under sedation, providing new anesthesia monitoring tools for clinical use.

DETAILED DESCRIPTION:
This is a single-center, prospective, observational clinical study. Study Objective: To explore the optimal sedation quality for painless gastrointestinal endoscopy. Study Protocol: A total of 220 patients undergoing painless gastrointestinal endoscopy were selected, with 110 patients undergoing gastroscopy and 110 patients undergoing colonoscopy. The bispectral index monitor (Apollo-9000A) was used to monitor the qCON and qNOX values of patients during the painless gastrointestinal endoscopy. The changes in qCON, qNOX, SBP (systolic blood pressure), DBP (diastolic blood pressure), MAP (mean arterial pressure), HR (heart rate), SpO2 (peripheral capillary oxygen saturation), and MOAA/S (Modified Observer's Assessment of Alertness/Sedation) scores at different time points during gastroscopy and colonoscopy were observed and recorded. The occurrence of adverse events during and after the examinations was also documented.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-60 years old;
2. American Society of Anesthesiologists (ASA) Class I-III;
3. Body mass index (BMI): 18-30 kg/m^2;
4. Individuals scheduled for elective gastroscopy and colonoscopy examinations;
5. Willing to comply with the experimental procedures and voluntarily sign the informed consent form

Exclusion Criteria:

1. Pregnant or breastfeeding women;
2. Individuals with allergies to sedatives/anesthetic drugs or other severe anesthetic risks;
3. Patients with chronic preoperative pain or a history of substance abuse;
4. Individuals with severe neurological diseases, such as stroke, hemiplegia, seizures, epilepsy, etc.;
5. Patients with clearly difficult airways, such as those with limited mouth opening, neck or jaw mobility restrictions, rheumatoid arthritis, or temporomandibular joint disorders;
6. Individuals with respiratory diseases, such as bronchitis, asthma, chronic obstructive pulmonary disease, or acute respiratory infections, which may lead to increased airway sensitivity;
7. Patients with chronic pharyngitis, laryngitis, laryngeal edema, or recurrent laryngeal nerve paralysis that may affect normal throat function;
8. Individuals with esophagitis, esophageal strictures, or esophageal motility disorders that may cause difficulty swallowing or reflux;
9. Patients with poorly controlled life-threatening cardiovascular diseases, such as uncontrolled severe hypertension, severe arrhythmias, or unstable angina; 10.10.Patients with liver dysfunction (Child-Pugh grade C or above), acute upper gastrointestinal bleeding with shock, severe anemia, or gastrointestinal obstruction with retained gastric contents.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Aged 18-60 years old;Individuals scheduled for elective gastroscopy and colonoscopy examinations
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Anesthesia quality | during the procedure
  The quality of anesthesia and sedation during gastroscopy through the throat or colonoscopy through the anus (criteria: HR and SBP fluctuations within 10%; no movement or coughing response)

SECONDARY OUTCOMES:
The values of qCON 、 qNOX、MAP、HR、SPO2 、and MOAA/S at different time points | during the procedure
  The Values of qCON 、 qNOX、MAP、HR、SPO2 and MOAA/S at different time points during gastroscopy and enteroscopy ① Time points for gastroscopy: Baseline value (T0), Loss of consciousness (T1), Before insertion of the gastroscope (T2), Passage of the gastroscope through the pharynx (T3), After insertion of the gastroscope (T4), Withdrawal of the gastroscope to the pharynx (T5), Examination completion (T6), Admission to recovery room (T7), Awakening (T8), Discharge from recovery room (T9).
  ② Time points for colonoscopy: Baseline value (T0), Loss of consciousness (T1), Before insertion of the colonoscope (T2), After insertion of the colonoscope into the anus (S3), Descending colon (T4), Splenic flexure (T5), Hepatic flexure (T6), Examination completion (T7), Admission to recovery room (T8), Awakening (T9), Discharge from recovery room (T10).
The values of qCON 、 qNOX、MAP、HR、SPO2 under special events | during the procedure
  During gastroscopy and colonoscopy , the values of qCON 、 qNOX、MAP、HR、SPO2 are recorded when coughing, body movement, polypectomy, or biopsy occur.
Adverse event | during the procedure
  Adverse events during gastroscopy and enteroscopy were recorded, including hypotension, hypertension, tachycardia, bradycardia, respiratory depression, hypoxemia, cough, body movement, nausea, vomiting, hiccup, injection pain, abdominal pain, abdominal distension, reflux aspiration.
Adverse events and complications after examination | 24 hours after procedure
  Bleeding, dizziness, blurred vision, nausea, vomiting, abdominal pain, abdominal distension were followed up 24h after the examination

CONTACTS AND LOCATIONS:
Overall Officials: Su Min, Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- China,Chongqing The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China